CLINICAL TRIAL: NCT02875769
Title: Effectiveness of a Pre-procedural Mouthwash in Reducing Bacteria in Dental Aerosols and Splatters: a Randomized Clinical Trial
Brief Title: Pre-procedural Mouthwash in Reducing Bacteria in Dental Aerosols
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Belén Retamal-Valdes, DDS, MSc, PhD Student, University of Guarulhos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAAE: 41244315.4.0000.5506
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Chronic Periodontitis
Keywords: cetylpyridinium chloride; chlorhexidine; oral aerosol; oral splatter; mouthwash; microbiology
MeSH Terms: conditions — Chronic Periodontitis | interventions — Dental Prophylaxis; Water

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test: Mouthwash CPC+Zn+F (Experimental): To rinse with pre-procedural mouthwash containing 0.075% cetylpyridinium chloride, 0.28% zinc lactate and 0.05% sodium fluoride in an Alcohol-free base (for one minute and 20 ml of solution) + full mouth dental prophylaxis using ultrasonic scaler.
  Interventions: Procedure: Dental prophylaxis; Drug: Mouthwash CPC+Zn+F
- Positive control: Mouthwash CHX (Active Comparator): To rinse with pre-procedural mouthwash containing 0.12% CHX with 10% alcohol (for one minute and 20 ml of solution) + full mouth dental prophylaxis using ultrasonic scaler.
  Interventions: Procedure: Dental prophylaxis; Drug: Mouthwash CHX
- Negative control A: No rinsing (Placebo Comparator): No rinsing with pre-procedural mouthwash + full mouth dental prophylaxis using ultrasonic scaler.
  Interventions: Procedure: Dental prophylaxis; Other: No rinsing
- Negative control B: Water (Placebo Comparator): To rinse with pre-procedural mouthwash containing water from a three-way syringe (for one minute and 20 ml of solution) + full mouth dental prophylaxis using ultrasonic scaler.
  Interventions: Procedure: Dental prophylaxis; Other: Water

INTERVENTIONS:
Procedure: Dental prophylaxis — Full mouth dental prophylaxis (FMDP) was conducted in one appointment lasting 10 minute, using an ultrasonic scaler at a frequency of 25 kHz (Cavitron Select SPC, Dentsply professional, York, PA, USA) at less than 50% power. The FMDP performed without anesthesia and in order to eliminate supragingival plaque, calculus and stainings.
Drug: Mouthwash CPC+Zn+F — The volunteer rinsed with pre-procedural mouthwash containing 0.075% cetylpyridinium chloride, 0.28% zinc lactate and 0.05% sodium fluoride in an Alcohol-free base for one minute, 20 ml of solution and then expectorated all remaining liquid.
  Other Names: Pre-procedural mouthwash CPC+Zn+F
  Arms: Test: Mouthwash CPC+Zn+F
Drug: Mouthwash CHX — The volunteer rinsed with pre-procedural mouthwash containing 0.12% CHX with 10% alcohol for one minute, 20 ml of solution and then expectorated all remaining liquid.
  Other Names: Pre-procedural mouthwash
  Arms: Positive control: Mouthwash CHX
Other: No rinsing — The volunteer did not rinse with any pre-procedural mothwash.
  Arms: Negative control A: No rinsing
Other: Water — The volunteer rinsed with pre-procedural mouthwash containing water from a three-way syringe for one minute, 20 ml of water and then expectorated all remaining liquid.
  Arms: Negative control B: Water

SUMMARY:
The aim of this randomized, single blinded clinical trial was to evaluate the effect of a pre-procedural mouthwash containing cetylpyridinium chloride (CPC), zinc lactate (Zn) and sodium fluoride (F) in the reduction of viable bacteria in oral aerosol/splatter after a dental prophylaxis with ultrasonic scaler.

DETAILED DESCRIPTION:
The propagation of oral microorganisms in the dental office during different oral procedures has been a concern. The use of certain equipment such as ultrasonic devices, highspeed dental handpieces or three-way syringes may spread aerosols and splatters containing microorganisms in the environment. These microorganisms may cause cross-infections in the dental office, jeopardizing the health of patients and dental professionals. Different procedures, materials and antimicrobial agents have been proposed to minimize microbial cross-contamination in the dental office. Chlorhexidine (CHX) is considered the gold standard substance in controlling oral biofilm growth in the oral cavity or microbial spread by oral aerosols due to its broad antibacterial spectrum and substantivity of 8 to 12 hours. However, other antiseptics have also been used as pre-procedural mouthwashes. CPC has an important antimicrobial activity and is considered a safe product for marketing. In this context, the present trend has been to combine more than one active substance in mouthwash and toothpaste formulations with the aim of increasing the efficacy of the products, or treating more than one clinical problem, such as plaque accumulation and halitosis, caries or gingival inflammation. Therefore, the aim of this randomized clinical trial (RCT) was to evaluate the effectiveness of a new mouthwash formulation containing 0.075% CPC, 0.28% zinc lactate and 0.05% sodium fluoride (CPC+Zn+F) in reducing viable bacteria present in oral aerosol/splatter. Sixty systemically healthy volunteers receiving dental prophylaxis were randomly assigned to one of the following experimental groups (15 per group): i) rinsing with 0.075% CPC, 0.28% Zn and 0.05% F (CPC+Zn+F), ii) 0.12% chlorhexidine digluconate (CHX), iii) no rinsing and iv) rinsing with water. Viable bacteria were collected from different locations in the dental office on enriched TSA plates and anaerobically incubated for 72 hours. The colonies were counted and species were then identified by Checkerboard DNA-DNA Hybridization. The total number of colony-forming units (CFUs) detected in the aerosols/splatters from volunteers who rinsed with CPC+Zn+F or CHX was statistically significantly (p<0.05) lower than of those subjects who did not rinse or who rinsed with water. When all locations were considered together, the aerosols/splatters from the CPC+Zn+F and CHX groups showed, respectively, 70% and 77% fewer CFUs than those from the no rinsing group and 61% and 70% than those from the water group. The mean proportions of bacterial species from the orange complex were statistically significantly (p<0.05) lower in aerosols/splatter from the CPC+Zn+F and CHX groups compared with the two negative controls. In conclusion, the results of the present investigation showed that a mouthwash containing 0.075% CPC, 0.28% Zn and 0.05% F, is effective in reducing viable bacteria in oral aerosol/splatter after a dental prophylaxis with ultrasonic scaler. This finding is highly relevant to the clinical practice, as it may greatly reduce the risk of cross-contamination in dental offices.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years;
* minimum of 20 natural teeth (excluding third molars and teeth with advanced decay indicated for extraction);
* at least 80% of the sites with visible supragingival plaque;
* fewer than 10% of sites with visible supragingival calculus;
* fewer than 30% of sites with probing depth (PD) ≥ 5 mm.

Exclusion Criteria:

* presence of orthodontic bands;
* partial removable dentures;
* lesions of the soft or hard tissues of the oral cavity;
* carious lesions requiring immediate restorative treatment;
* history of allergy to CHX, CPC, zinc lactate or sodium fluoride;
* participation in any other clinical study within the one-month period prior to entering into the study;
* professional tooth cleaning procedure (oral prophylaxis) during the period of one month prior to entering the study;
* pregnant or breast-feeding women;
* antibiotic therapy in the previous 6 months;
* continuous use of oral mouthwashes;
* any systemic condition that may require prophylactic medication for dental treatment (e.g., mitral valve prolapse).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Difference between groups (test, positive control, negative control A and negative control B) for the mean number of total colony-forming units (CFUs) in all plates. | During oral prophylaxis procedure.

SECONDARY OUTCOMES:
Number of total CFUs in plates positioned on the clinician forehead. | During oral prophylaxis procedure.
Number of total CFUs in plates positioned on the volunteer's chest. | During oral prophylaxis procedure.
Number of total CFUs in plates positioned on the support board. | During oral prophylaxis procedure.
Proportion of the microbial complexes. | During oral prophylaxis procedure.
Reduction in CFUs in the CPC+Zn+F and CHX groups in comparison with the two negative control groups. | During oral prophylaxis procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Feres, Professor, Study Chair — Guarulhos University

IPD SHARING:
Plan to Share IPD: Yes
September 2016

REFERENCES:
- [Background] Bentley CD, Burkhart NW, Crawford JJ. Evaluating spatter and aerosol contamination during dental procedures. J Am Dent Assoc. 1994 May;125(5):579-84. doi: 10.14219/jada.archive.1994.0093. PMID 8195499
- [Background] Cochran MA, Miller CH, Sheldrake MA. The efficacy of the rubber dam as a barrier to the spread of microorganisms during dental treatment. J Am Dent Assoc. 1989 Jul;119(1):141-4. doi: 10.14219/jada.archive.1989.0131. PMID 2760346
- [Background] Erovic Ademovski S, Lingstrom P, Renvert S. The effect of different mouth rinse products on intra-oral halitosis. Int J Dent Hyg. 2016 May;14(2):117-23. doi: 10.1111/idh.12148. Epub 2015 May 31. PMID 26031397
- [Background] Grenier D. Quantitative analysis of bacterial aerosols in two different dental clinic environments. Appl Environ Microbiol. 1995 Aug;61(8):3165-8. doi: 10.1128/aem.61.8.3165-3168.1995. PMID 7487047
- [Background] Gupta G, Mitra D, Ashok KP, Gupta A, Soni S, Ahmed S, Arya A. Efficacy of preprocedural mouth rinsing in reducing aerosol contamination produced by ultrasonic scaler: a pilot study. J Periodontol. 2014 Apr;85(4):562-8. doi: 10.1902/jop.2013.120616. Epub 2013 Jul 15. PMID 23855840
- [Background] Harrel SK, Molinari J. Aerosols and splatter in dentistry: a brief review of the literature and infection control implications. J Am Dent Assoc. 2004 Apr;135(4):429-37. doi: 10.14219/jada.archive.2004.0207. PMID 15127864
- [Background] Jones CG. Chlorhexidine: is it still the gold standard? Periodontol 2000. 1997 Oct;15:55-62. doi: 10.1111/j.1600-0757.1997.tb00105.x. PMID 9643233
- [Background] Kanjirath PP, Coplen AE, Chapman JC, Peters MC, Inglehart MR. Effectiveness of gloves and infection control in dentistry: student and provider perspectives. J Dent Educ. 2009 May;73(5):571-80. PMID 19433532
- [Background] Keni NN, Aras MA, Chitre V. Chlorhexidine allergy due to topical application. Indian J Dent Res. 2012 Sep-Oct;23(5):674-6. doi: 10.4103/0970-9290.107393. PMID 23422617
- [Background] Kjaerheim V, Skaare A, Barkvoll P, Rolla G. Antiplaque, antibacterial, and anti-inflammatory properties of triclosan mouthrinses in combination with zinc citrate or polyvinylmethylether maleic acid (PVM-MA) copolymer. Eur J Oral Sci. 1996 Oct-Dec;104(5-6):529-34. doi: 10.1111/j.1600-0722.1996.tb00137.x. PMID 9021321
- [Background] Lang C, Murgia C, Leong M, Tan LW, Perozzi G, Knight D, Ruffin R, Zalewski P. Anti-inflammatory effects of zinc and alterations in zinc transporter mRNA in mouse models of allergic inflammation. Am J Physiol Lung Cell Mol Physiol. 2007 Feb;292(2):L577-84. doi: 10.1152/ajplung.00280.2006. Epub 2006 Nov 3. PMID 17085522
- [Background] Leggat PA, Kedjarune U. Bacterial aerosols in the dental clinic: a review. Int Dent J. 2001 Feb;51(1):39-44. doi: 10.1002/j.1875-595x.2001.tb00816.x. PMID 11326448
- [Background] Legnani P, Checchi L, Pelliccioni GA, D'Achille C. Atmospheric contamination during dental procedures. Quintessence Int. 1994 Jun;25(6):435-9. PMID 7938434
- [Background] Mendes L, Coimbra J, Pereira AL, Resende M, Pinto MG. Comparative effect of a new mouthrinse containing chlorhexidine, triclosan and zinc on volatile sulphur compounds: a randomized, crossover, double-blind study. Int J Dent Hyg. 2016 Aug;14(3):202-8. doi: 10.1111/idh.12132. Epub 2015 Feb 26. PMID 25727335
- [Background] Nejatidanesh F, Khosravi Z, Goroohi H, Badrian H, Savabi O. Risk of Contamination of Different Areas of Dentist's Face During Dental Practices. Int J Prev Med. 2013 May;4(5):611-5. PMID 23930175
- [Background] Pandit S, Cai JN, Jung JE, Lee YS, Jeon JG. Effect of brief cetylpyridinium chloride treatments during early and mature cariogenic biofilm formation. Oral Dis. 2015 Jul;21(5):565-71. doi: 10.1111/odi.12312. Epub 2015 Feb 13. PMID 25600577
- [Background] Rivera-Hidalgo F, Barnes JB, Harrel SK. Aerosol and splatter production by focused spray and standard ultrasonic inserts. J Periodontol. 1999 May;70(5):473-7. doi: 10.1902/jop.1999.70.5.473. PMID 10368050
- [Background] Slots J. Low-cost periodontal therapy. Periodontol 2000. 2012 Oct;60(1):110-37. doi: 10.1111/j.1600-0757.2011.00429.x. PMID 22909110
- [Background] Socransky SS, Haffajee AD, Cugini MA, Smith C, Kent RL Jr. Microbial complexes in subgingival plaque. J Clin Periodontol. 1998 Feb;25(2):134-44. doi: 10.1111/j.1600-051x.1998.tb02419.x. PMID 9495612
- [Background] Souza-Gugelmin MC, Lima CD, Lima SN, Mian H, Ito IY. Microbial contamination in dental unit waterlines. Braz Dent J. 2003;14(1):55-7. doi: 10.1590/s0103-64402003000100010. Epub 2003 Jul 31. PMID 12656466
- [Background] Thomas E. Efficacy of two commonly available mouth rinses used as preprocedural rinses in children. J Indian Soc Pedod Prev Dent. 2011 Apr-Jun;29(2):113-6. doi: 10.4103/0970-4388.84682. PMID 21911948
- [Background] Timmerman MF, Menso L, Steinfort J, van Winkelhoff AJ, van der Weijden GA. Atmospheric contamination during ultrasonic scaling. J Clin Periodontol. 2004 Jun;31(6):458-62. doi: 10.1111/j.1600-051X.2004.00511.x. PMID 15142216
- [Background] Toroglu MS, Haytac MC, Koksal F. Evaluation of aerosol contamination during debonding procedures. Angle Orthod. 2001 Aug;71(4):299-306. doi: 10.1043/0003-3219(2001)0712.0.CO;2. PMID 11510639
- [Background] Varoni E, Tarce M, Lodi G, Carrassi A. Chlorhexidine (CHX) in dentistry: state of the art. Minerva Stomatol. 2012 Sep;61(9):399-419. English, Italian. PMID 22976567
- [Background] Veena HR, Mahantesha S, Joseph PA, Patil SR, Patil SH. Dissemination of aerosol and splatter during ultrasonic scaling: a pilot study. J Infect Public Health. 2015 May-Jun;8(3):260-5. doi: 10.1016/j.jiph.2014.11.004. Epub 2015 Jan 3. PMID 25564419
- [Background] Yengopal V. The use of essential oil mouthwashes as preprocedural rinses for infection control. SADJ. 2004 Jul;59(6):247-8, 250. No abstract available. PMID 15457911
- [Result] Costa X, Laguna E, Herrera D, Serrano J, Alonso B, Sanz M. Efficacy of a new mouth rinse formulation based on 0.07% cetylpyridinium chloride in the control of plaque and gingivitis: a 6-month randomized clinical trial. J Clin Periodontol. 2013 Nov;40(11):1007-15. doi: 10.1111/jcpe.12158. Epub 2013 Sep 11. PMID 24024983
- [Result] Feres M, Figueiredo LC, Faveri M, Stewart B, de Vizio W. The effectiveness of a preprocedural mouthrinse containing cetylpyridinium chloride in reducing bacteria in the dental office. J Am Dent Assoc. 2010 Apr;141(4):415-22. doi: 10.14219/jada.archive.2010.0193. PMID 20354090
- [Result] Giertsen E. Effects of mouthrinses with triclosan, zinc ions, copolymer, and sodium lauryl sulphate combined with fluoride on acid formation by dental plaque in vivo. Caries Res. 2004 Sep-Oct;38(5):430-5. doi: 10.1159/000079623. PMID 15316186
- [Result] Kang JH, Jang YJ, Kim DJ, Park JW. Antimicrobial effectiveness of cetylpyridinium chloride and zinc chloride-containing mouthrinses on bacteria of halitosis and peri-implant disease. Int J Oral Maxillofac Implants. 2015 Nov-Dec;30(6):1341-7. doi: 10.11607/jomi.3824. Epub 2015 Oct 16. PMID 26478974
- [Result] Kaur R, Singh I, Vandana KL, Desai R. Effect of chlorhexidine, povidone iodine, and ozone on microorganisms in dental aerosols: randomized double-blind clinical trial. Indian J Dent Res. 2014 Mar-Apr;25(2):160-5. doi: 10.4103/0970-9290.135910. PMID 24992844
- [Result] Logothetis DD, Martinez-Welles JM. Reducing bacterial aerosol contamination with a chlorhexidine gluconate pre-rinse. J Am Dent Assoc. 1995 Dec;126(12):1634-9. doi: 10.14219/jada.archive.1995.0111. PMID 7499664
- [Result] Reddy S, Prasad MG, Kaul S, Satish K, Kakarala S, Bhowmik N. Efficacy of 0.2% tempered chlorhexidine as a pre-procedural mouth rinse: A clinical study. J Indian Soc Periodontol. 2012 Apr;16(2):213-7. doi: 10.4103/0972-124X.99264. PMID 23055587
- [Result] Shetty SK, Sharath K, Shenoy S, Sreekumar C, Shetty RN, Biju T. Compare the effcacy of two commercially available mouthrinses in reducing viable bacterial count in dental aerosol produced during ultrasonic scaling when used as a preprocedural rinse. J Contemp Dent Pract. 2013 Sep 1;14(5):848-51. doi: 10.5005/jp-journals-10024-1414. PMID 24685786

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02875769/SAP_000.pdf